CLINICAL TRIAL: NCT06059846
Title: A Phase 3, Randomized, Double-blind, Double-dummy, Multicenter, Multinational Study to Assess the Efficacy and Safety of Orally Administered Tebipenem Pivoxil Hydrobromide (TBP-PI-HBr) Compared to Intravenously Administered Imipenem-cilastatin in Patients With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Brief Title: A Study of Oral Tebipenem Pivoxil Hydrobromide (TBP-PI-HBr) Compared to Intravenous Imipenem-cilastatin in Participants With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Acronym: PIVOT-PO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPR994-305; 2023-503785-22-00 (Other: EU CT Number)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections | interventions — tebipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TBP-PI-HBr 600 mg + Dummy Infusion (Experimental): Participants will receive TBP-PI-HBr 600 mg, orally and dummy infusion IV, every 6 hours from Days 1 through 10.
  Interventions: Drug: TBP-PI-HBr; Drug: Dummy Infusion
- Imipenem-cilastatin 500 mg + Dummy Tablets (Active Comparator): Participants will receive imipenem-cilastatin 500 mg, IV and matched dummy tablets, orally, every 6 hours from Days 1 through 10.
  Interventions: Drug: Imipenem-cilastatin; Drug: Dummy Tablets

INTERVENTIONS:
Drug: TBP-PI-HBr — TBP-PI-HBr film-coated immediate-release tablets.
  Other Names: SPR994
  Arms: TBP-PI-HBr 600 mg + Dummy Infusion
Drug: Imipenem-cilastatin — Sterile powder for reconstitution administered as IV.
  Arms: Imipenem-cilastatin 500 mg + Dummy Tablets
Drug: Dummy Infusion — 0.9% sodium chloride administered as IV infusion.
  Arms: TBP-PI-HBr 600 mg + Dummy Infusion
Drug: Dummy Tablets — TBP-PI-HBr matching dummy tablets.
  Arms: Imipenem-cilastatin 500 mg + Dummy Tablets

SUMMARY:
The primary purpose of this study is to assess the efficacy of oral TBP-PI-HBr as compared with intravenous (IV) imipenem-cilastatin with respect to the overall response (combined clinical cure plus microbiological eradication) at the Test-of-Cure (TOC) visit in hospitalized adult participants (≥18 years of age) with cUTI or AP.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of cUTI or AP.
2. Have an adequate urine specimen for evaluation and culture obtained within 24 hours prior to randomization with evidence of pyuria that includes at least one of the following:

   1. at least 10 white blood cells (WBCs) per high power field (HPF) in urine sediment
   2. at least 10 WBCs per millimeters cubed (mm^3) in unspun urine
   3. positive leukocyte esterase (LE) on urinalysis Note: Participants may be randomized and administered study drug prior to knowledge of urine culture results, but pyuria must be documented.
3. Expectation, in the judgment of the Investigator, that the participant will survive with effective antimicrobial therapy and appropriate supportive care for the anticipated duration of the study.

Exclusion Criteria:

1. Presence of any known or suspected disease or condition that may confound the assessment of efficacy.
2. Gross hematuria requiring intervention other than administration of study drug or removal/placement of urinary tract instrumentation.
3. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period.
4. Creatinine clearance (CrCl) of ≤30 milliliters per minute (mL/min), as estimated by the Cockcroft-Gault formula.
5. Anticipated concomitant use of non-study antimicrobial drug therapy between randomization and the LFU visit that would potentially effect outcome evaluations of cUTI/AP.
6. Receipt of a potentially effective antimicrobial within 72 hours prior to study randomization.
7. Severe hepatic impairment at Screening, as evidenced by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5×upper limit of normal (ULN) or total bilirubin >3×ULN, or clinical signs of cirrhosis or end-stage hepatic disease (e.g., ascites, hepatic encephalopathy).
8. Pregnant or lactating women.
9. History of epilepsy or known seizure disorder (excluding a history of childhood febrile seizures).
10. History of proven or suspected Clostridioides difficile associated diarrhea.
11. History of human immunodeficiency virus (HIV) infection.
12. QT interval corrected using Fridericia's formula (QTcF) >480 milliseconds (msec) based on screening ECG.
13. History of known genetic metabolism anomaly associated with carnitine deficiency.
14. Requirement for concomitant use of valproic acid, divalproex sodium, or probenecid between randomization and EOT.

Note: Other inclusion and exclusion criteria as per protocol may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1690 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Overall Response at the Test-of-Cure (TOC) Visit | Day 17
  Overall response includes combination of clinical cure and favorable microbiological response. Clinical cure is defined as a complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at Baseline and no new symptoms, such that no further antibacterial therapy is warranted, and participant is alive. Favorable microbiological response (microbiological eradication) is defined as a reduction of Baseline uropathogens to <10^3 colony forming unit per milliliter (CFU/mL) and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline and participant is alive.

SECONDARY OUTCOMES:
Number of Participants in the Microbiologically Evaluable Population With Overall Response at the TOC Visit | Day 17
  Overall response includes combination of clinical cure and favorable microbiological response. Clinical cure is defined as a complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at Baseline and no new symptoms, such that no further antibacterial therapy is warranted, and participant is alive. Favorable microbiological response (microbiological eradication) is defined as a reduction of Baseline uropathogens to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at Baseline and participant is alive.
Number of Participants With Overall Response at the End-of-Treatment (EOT) and Late Follow-Up (LFU) Visits | Days 10 and 28
  Overall response includes combination of clinical cure and favorable microbiological response. Clinical cure is defined as a complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at Baseline and no new symptoms, such that no further antibacterial therapy is warranted, and participant is alive. Favorable microbiological response (microbiological eradication) is defined as a reduction of Baseline uropathogens to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at Baseline and participant is alive.
Number of Participants With Clinical Response at the EOT, TOC and LFU Visits | Days 10, 17, and 28
  Participants will be evaluated for clinical response outcome based on assessment of signs and symptoms as: Cure, including sustained clinical cure: Sustained clinical cure is defined as met criteria for clinical cure at TOC, and remained free of new or recurrent signs and symptoms of cUTI or AP at LFU visit such that no further antibacterial therapy is warranted; Failure, including clinical relapse: Clinical relapse is defined as met criteria for clinical cure at TOC, but new signs and symptoms of cUTI or AP are present at LFU visit and participant requires antibacterial therapy for cUTI; Clinical indeterminate: insufficient data are available to determine if participant is a sustained clinical cure or clinical relapse. If a participant is assessed as a clinical failure at EOT, participant is automatically considered a failure at TOC and LFU visits. If a participant is assessed as a clinical failure at TOC, participant is automatically considered a failure at LFU visit.
Number of Participants With Microbiological Response at the EOT, TOC and LFU Visits | Days 10, 17, and 28
  Participants will be evaluated for microbiological response based on blood and urine cultures as:Eradication, including sustained microbiologic eradication, i.e.,microbiologic eradication at TOC and no subsequent urine culture after TOC demonstrating recurrence of original Baseline uropathogen at ≥10^3 CFU/mL;Persistence, including microbiologic recurrence, i.e.,isolation from urine culture at ≥10^3 CFU/mL or blood culture of any of Baseline uropathogen(s) at any time after documented eradication at TOC visit up to and including LFU visit;Microbiologic indeterminate:no follow-up urine culture is available, or urine culture results are missing, or follow-up urine culture cannot be interpreted for any reason. If a participant is assessed as a microbiological persistence at EOT,participant is automatically considered persistent at TOC and LFU. If assessed as persistent at TOC, participant is automatically considered a persistent at LFU.
Number of Participants With Overall Response at the EOT, TOC, and LFU Visits in Participants With Drug-resistant Enterobacterales | Days 10, 17, and 28
  Overall response includes combination of clinical cure and favorable microbiological response. Clinical cure is defined as a complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at Baseline and no new symptoms, such that no further antibacterial therapy is warranted, and participant is alive. Favorable microbiological response (microbiological eradication) is defined as a reduction of Baseline uropathogens to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at Baseline and participant is alive.
Number of Participants With Clinical Response at the EOT, TOC, and LFU Visits in Participants With Drug-resistant Enterobacterales | Days 10, 17, and 28
  Participants will be evaluated for clinical response outcome based on assessment of signs and symptoms as: Cure, including sustained clinical cure: Sustained clinical cure is defined as met criteria for clinical cure at TOC, and remained free of new or recurrent signs and symptoms of cUTI or AP at LFU visit such that no further antibacterial therapy is warranted; Failure, including clinical relapse: Clinical relapse is defined as met criteria for clinical cure at TOC, but new signs and symptoms of cUTI or AP are present at LFU visit and participant requires antibacterial therapy for cUTI; Clinical indeterminate: insufficient data are available to determine if participant is a sustained clinical cure or clinical relapse. If a participant is assessed as a clinical failure at EOT, participant is automatically considered a failure at TOC and LFU visits. If a participant is assessed as a clinical failure at TOC, participant is automatically considered a failure at LFU visit.
Number of Participants With Microbiological Response at the EOT, TOC, and LFU Visits in Participants With Drug-resistant Enterobacterales | Days 10, 17, and 28
  Participants will be evaluated for microbiological response based on blood and urine cultures as:Eradication, including sustained microbiologic eradication, i.e.,microbiologic eradication at TOC and no subsequent urine culture after TOC demonstrating recurrence of original Baseline uropathogen at ≥10^3 CFU/mL;Persistence, including microbiologic recurrence, i.e.,isolation from urine culture at ≥10^3 CFU/mL or blood culture of any of Baseline uropathogen(s) at any time after documented eradication at TOC visit up to and including LFU visit;Microbiologic indeterminate:no follow-up urine culture is available, or urine culture results are missing, or follow-up urine culture cannot be interpreted for any reason. If a participant is assessed as a microbiological persistence at EOT,participant is automatically considered persistent at TOC and LFU. If assessed as persistent at TOC, participant is automatically considered a persistent at LFU.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first dose of study drug (Day 1) up to Day 28
Plasma Concentration of Tebipenem | At multiple time points post dose on Day 2

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Study Director — Spero Therapeutics
Locations (84):
- United States (2):
  - Medical facility, Miami, Florida
  - Medical Facility, Miami, Florida
- Argentina (6):
  - Medical Facility, Buenos Aires
  - Medical Facility, Córdoba
  - Medical Facility, La Plata
  - Medical Facility, Mendoza
  - Medical Facility, San Miguel de Tucumán
  - Medical Facility, Villa Regina
- Bosnia and Herzegovina (3):
  - Medical Facility, Banja Luka
  - Medical Facility, Sarajevo
  - Medical Facility, Tuzla
- Brazil (5):
  - Medical Facility, Barueri
  - Medical Facility, Campinas
  - Medical Facility, Curitiba
  - Medical Facility, Porto Alegre
  - Medical Facility, São José do Rio Preto
- Bulgaria (11):
  - Medical Facility, Blagoevgrad
  - Medical Facility, Dobrich
  - Medical Facility, Gabrovo
  - Medical facility, Lom
  - Medical Facility, Pleven
  - Medical Facility, Plovdiv
  - Medical facility, Rousse
  - Medical facility, Shumen
  - Medical Facility, Sliven
  - Medical facility, Sofia
  - Medical Facility, Varna
- Croatia (4):
  - Medical Facility, Čakovec
  - Medical Facility, Slavonski Brod
  - Medical Facility, Split
  - Medical Facility, Zagreb
- Estonia (4):
  - Medical Facility, Kohtla-Järve
  - Medical Facility, Pärnu
  - Medical Facility, Tallinn
  - Medical Facility, Võru
- Medical facility, Tbilisi, Georgia
- Greece (5):
  - Medical Facility, Alexandroupoli
  - Medical Facility, Athens
  - Medical Facility, Ioannina
  - Medical Facility, Pátrai
  - Medical Facility, Thessaloniki
- Hungary (4):
  - Medical Facility, Budapest
  - Medical Facility, Eger
  - Medical Facility, Kistarcsa
  - Medical Facility, Nyíregyháza
- India (5):
  - Medical Facility, Varanasi, Uttar Pradesh
  - Medical Facility, Bangalore
  - Medical Facility, Belagavi
  - Medical Facility, Jaipur
  - Medical Facility, Lucknow
- Latvia (4):
  - Medical Facility, Daugavpils
  - Medical Facility, Liepāja
  - Medical Facility, Riga
  - Medical Facility, Valmiera
- Medical Facility, Chisinau, Moldova
- Poland (4):
  - Medical Facility, Krakow
  - Medical Facility, Lodz
  - Medical Facility, Warsaw
  - Medical Facility, Łęczna
- Romania (6):
  - Medical Facility, Brasov
  - Medical facility, Bucharest
  - Medical facility, Craiova
  - Medical Facility, Iași
  - Medical Facility, Oradea
  - Medical Facility, Timișoara
- Serbia (4):
  - Medical facility, Belgrade
  - Medical facility, Kragujevac
  - Medical facility, Niš
  - Medical facility, Novi Sad
- Slovakia (5):
  - Medical Facility, Bratislava
  - Medical Facility, Galanta
  - Medical Facility, Lučenec
  - Medical Facility, Malacky
  - Medical Facility, Poprad
- South Africa (5):
  - Medical facility, Benoni
  - Medical facility, Durban
  - Medical Facility, Pretoria
  - Medical Facility, Tongaat
  - Medical Facility, Umhlanga
- Turkey (Türkiye) (5):
  - Medical Facility, Ankara
  - Medical Facility, Diyarbakır
  - Medical Facility, Istanbul
  - Medical Facility, Izmir
  - Medical Facility, Samsun

IPD SHARING:
Plan to Share IPD: No